CLINICAL TRIAL: NCT06549114
Title: A Study to Assess Safety and Tolerability, and Explore Efficacy of Leniolisib for Immune Dysregulation in Primary Immunodeficiency Disorders
Brief Title: Leniolisib for Immune Dysregulation in PIDs
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pharming Technologies B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LE 7201
Record Dates: First submitted 2024-07-17; First posted 2024-08-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Primary Immunodeficiency Disorders (PIDs)
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — leniolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Leniolisib (Experimental): All subjects participating will receive Leniolisib film-coated tablets (FCTs) at a starting dose of 10 mg BID for 4 weeks, followed by 30 mg BID for 4 weeks, and then 70 mg BID for 12 weeks.
  Interventions: Drug: Leniolisib

INTERVENTIONS:
Drug: Leniolisib — The doses selected will range from 10 to 70 mg twice daily (BID) (resulting in total daily doses ranging from 20 to 140 mg per day).
  Other Names: Joenja

SUMMARY:
This study is an exploratory, non-randomized, open-label, within-patient dose escalation study. The primary objective is to assess safety and tolerability of leniolisib. Secondary objectives include assessments of PK/PD, and to explore clinical efficacy measures with administration of three different dose levels of leniolisib.

DETAILED DESCRIPTION:
Patients ages 12-75 diagnosed with genetically defined PID disorders linked to PI3K signaling. This includes disorders caused by pathogenic variants in SOCS1, PTEN, CTLA4, NFKB1 (variants leading to NFKB pathway activation), FAS (germline or somatic), or RAS-associated leukoproliferative disorder caused by somatic variants in NRAS or KRAS (not juvenile myelomonocytic leukemia [JMML]). All subjects participating will receive leniolisib film-coated tablets (FCTs) with a planned dose regimen consisting of a starting dose of 10 mg twice daily (BID) for 4 weeks, followed by 30 mg BID for 4 weeks, and then 70 mg BID for 12 weeks. Leniolisib dose increase at the individual subject level will occur if no safety or tolerability issues have been identified by the Investigator that precludes the planned dose escalation.

Subjects not continuing leniolisib treatment outside of the current protocol will be followed up, with the EOS visit planned to occur approximately 28 days after last dose of leniolisib.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 12 to 75 years of age.
2. Diagnosed with a PID due to disease-causing pathogenic or likely pathogenic variant(s) in the following genes: SOCS1, PTEN, CTLA4, NFKB1 (only those variants leading to NFKB pathway activation), or FAS (germline or somatic), or diagnosed with RAS associated leukoproliferative disorder (and not juvenile myelomonocytic leukemia [JMML]) due to somatic variants in NRAS or KRAS.
3. Subjects must have 1 or more of the following:

   * One or more blood cytopenias related to the underlying PID defined as hemoglobin <10 g/dL, platelet count <100,000/µL, or neutrophil count <1000/µL
   * Splenomegaly evident by CT imaging with craniocaudal spleen measurement >10 cm
   * Lymphadenopathy evident by CT imaging with at least 1 measurable index lymph node (long axis >1.5 cm) as per Cheson methodology
   * GLILD or other PID-related ILD with quantifiable CT chest imaging findings evident on baseline CT scan
4. At screening, vital signs.

   * Systolic blood pressure 80-139 mm Hg
   * Diastolic blood pressure 50-89 mm Hg
   * Pulse rate 50-110 bpm
   * Oxygen saturation 93-100%
5. Subjects or their legal representatives (for subjects under the age of 18 years) must be able to provide written informed consent.

Exclusion Criteria:

1. Subject has had a successful hematopoietic stem-cell transplant (HSCT).
2. Previous or concurrent use of immunosuppressive medication, such as:

   * Use of an mTOR inhibitor or a PI3Kδ inhibitor within 3 weeks prior to first dosing .
   * Rituximab or other B-cell depleting antibodies, belimumab, cyclophosphamide, or alemtuzumab within 6 months prior to first dosing.
   * Cyclosporine A, mycophenolate mofetil, 6-mercaptopurine, azathioprine, methotrexate, tacrolimus, ruxolitinib, or other JAK inhibitors within 3 weeks prior to first dosing.
   * Corticosteroids above 25 mg prednisone or equivalent per day within 2 weeks prior to first dosing.
   * Other immunosuppressive agents expected to have a significant impact on immune cell number or function.
   * Abatacept is allowed during study if the subject has been receiving a stable dosing regimen for more than 3 months prior to first dosing.
3. Subject is receiving concurrent treatment with another investigational therapy or use of another investigational therapy less than 4 weeks or 5 half-lives (whichever is longer) prior to first dosing.
4. History of hypersensitivity to the study drug or to drugs of similar chemical classes.
5. Current use of medication known to be a strong inhibitor, or moderate or strong inducer, of isoenzyme P450 CYP3A.
6. Current use of medications that act as BCRP, OATP1B1, and OATP1B3 substrates.
7. Subject has a history or current electrocardiogram (ECG) abnormalities indicating a significant risk of safety for subjects participating in the study
8. History of acquired immunodeficiency diseases, including a positive HIV test result at screening.
9. Uncontrolled chronic or recurrent infectious disease (except those considered to be characteristic of a PID) or evidence of tuberculosis infection
10. Any surgical or medical condition which may jeopardize the subject in case of participation in the study, or might significantly alter the absorption, distribution, metabolism, or excretion of drugs.
11. A positive hepatitis B surface antigen, positive hepatitis B PCR, positive hepatitis C PCR, or positive hepatitis C antibody result at screening.
12. Administration of live vaccines starting from 6 weeks before first dose of study medication.
13. Subject has a previous diagnosis of lymphoma within 1 year of the first dose of study medication.
14. Subject has a history of malignancy (except lymphoma) within 3 years before the first dose of study medication, except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.
15. Subject has uncontrolled post-transplant lymphoproliferative disease (PTLD)-like EBV related lymphoproliferative disease.
16. Donation or loss of 400 mL or more of blood within 8 weeks before the first dose.
17. Subject has had major surgery requiring hospitalization or radiotherapy within 4 weeks prior to the first dose or has a planned or expected major surgical procedure during the study period.
18. Pregnant or nursing (lactating) individuals,.
19. Individuals of child-bearing potential, unless they are using highly effective methods of contraception.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent adverse events (TEAEs), Serious Adverse Events (SAEs) , and Adverse Events (AEs) | From Baseline to the end of 20 weeks of Treatment
  • To assess the number of AEs/SAEs and number of participants with AEs/SAEs

SECONDARY OUTCOMES:
To assess the PK of leniolisib in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • PK parameters for leniolisib defined by Cmax
To assess the PK of leniolisib in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • PK parameters for leniolisib defined by Tmax
To assess the PK of leniolisib in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • PK parameters for leniolisib defined by t1/2
To assess the PK of leniolisib in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • PK parameters for leniolisib defined by AUC (0-t)
To assess the impact of leniolisib on lymphocyte PI3K/AKT/mTOR pathway activity in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • Percent change in pAKT and/or pS6 in B cells and/or T cells, under resting and stimulated conditions, at different dose levels of leniolisib relative to baseline pAKT/pS6 levels, as feasible
To assess the impact of leniolisib on hemoglobin counts in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • Hemoglobin over time
To assess the impact of leniolisib on platelet counts in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • Platelet count over time
To assess the impact of leniolisib on absolute neutrophil counts in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • Absolute neutrophil count over time
To assess the clinical efficacy of leniolisib on PID-related ILD in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • Change in CT evidence of GLILD or other PID-related ILD evaluated using Hartmann scoring methodology
To assess the clinical efficacy of leniolisib on PFTs in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • Change in forced expiratory volume 1 (FEV1)
To assess the clinical efficacy of leniolisib on PFTs in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • Change in forced vital capacity (FVC)
To assess the clinical efficacy of leniolisib on PFTs in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • Change in total lung capacity (TLC)
To assess the clinical efficacy of leniolisib on PFTs in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • Change in diffusing capacity (DLCO)
To assess the clinical efficacy of leniolisib on lymphoproliferation in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  * Percent change from baseline in lymphadenopathy measured as the sum of product of diameters (SPD) in the index lesions selected per the Cheson methodology
  * Percent change from baseline in lymphadenopathy measured as SPD of measurable non-index lesions selected as per the Cheson methodology
To assess the clinical efficacy of leniolisib on splenomegaly in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • Percent change from baseline in splenomegaly measured by three-dimensional (3D) volume and bi-dimensional (2D) size of spleen
To assess the impact of leniolisib on white blood cell counts in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • White blood cell count over time
To assess the impact of leniolisib on white blood cell counts in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • Absolute monocyte count over time
To assess the impact of leniolisib on white blood cell counts in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • Absolute lymphocyte count over time
To assess the impact of leniolisib on white blood cell counts in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • Absolute eosinophil count over time
To assess the impact of leniolisib on white blood cell counts in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • Absolute basophil count over time
To assess the impact of leniolisib on white blood cell counts in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • CD4+ T cell count over time
To assess the impact of leniolisib on white blood cell counts in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • CD8+ T cell count over time
To assess the impact of leniolisib on white blood cell counts in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • Natural killer (NK) cell count over time
To assess the impact of leniolisib on white blood cell counts in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • B cell count over time
To assess the impact of leniolisib on B cell and T cell phenotypic populations of interest in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  • Percentages of naïve B cells, CD21lo B cells and T regulatory cells over time
To examine levels of CXCL13 and soluble IL-2Rα and assess the impact of leniolisib in PID disorders linked to PI3K | From Baseline to the end of 20 weeks of Treatment
  * Levels of CXCL13 over time
  * Levels of soluble IL-2Rα over time

CONTACTS AND LOCATIONS:
Overall Officials: Gulbu Uzel, M.D., Principal Investigator — National Institutes of Health (NIH)
Locations (1):
- National Institute of Health, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hassan C, Ponstein Y, Hanssen R, Thorneloe KS, Marsh RA, Rao VK. Leniolisib reduced lymphoproliferative disease in murine autoimmune lymphoproliferative syndrome. J Hum Immun. 2025 Nov 17;2(1):e20250125. doi: 10.70962/jhi.20250125. eCollection 2026 Jan 5. PMID 41608120